CLINICAL TRIAL: NCT07057271
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial Designed to Evaluate the Efficacy and Safety of CJC-1134-PC Injection Administered Once A Week in Patients With Type 2 Diabetes With Inadequately Controlled Blood Glucose Level After Metformin Monotherapy or Metformin in Combination With Insulin Secretagogues
Brief Title: A Study of CJC-1134-PC Injection in Patients With Type 2 Diabetes With Inadequately Controlled Blood Glucose Level After Metformin Monotherapy or Metformin in Combination With Insulin Secretagogues
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changshan ConjuChem BioPharmaceutical Research and Development (Hebei) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSCJC DM301
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus - Poor Control

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CJC-1134-PC (Experimental): Injection, 0.2ml/2mg (prefilled pen)
  Interventions: Drug: CJC-1134-PC Injection
- Placebo (Placebo Comparator): Injection, 0.2ml/0mg (prefilled pen)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CJC-1134-PC Injection — Double-blind Treatment Period: 0.2ml (2mg) once weekly ×24 weeks (Week 1 to Week 24); Open-label Treatment Period: 0.2ml (2mg) once weekly ×28 weeks (Week 25 to Week 52)
  Arms: CJC-1134-PC
Drug: Placebo — Double-blind Treatment Period: 0.2ml (0mg) once weekly ×24 weeks (Week 1 to Week 24); Open-label Treatment Period: 0.2ml (2mg) once weekly ×28 weeks (Week 25 to Week 52)
  Arms: Placebo

SUMMARY:
This study is a Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial Designed to Evaluate the Efficacy and Safety of CJC-1134-PC Injection Administered Once A Week in Patients with Type 2 Diabetes with Inadequately Controlled Blood Glucose Level after Metformin Monotherapy or Metformin in Combination with Insulin Secretagogues.

ELIGIBILITY:
Inclusion Criteria:

Subjects were eligible for the study only if all the following inclusion criteria were met:

1. Males or females aged 18 - 70 years (inclusive) at screening;
2. Subjects with body mass index (BMI) ≥ 20 kg/ m2 and ≤ 40 kg/ m2.
3. Patients with type 2 diabetes diagnosed according to the World Health Organization (WHO) 1999 criteria and who have received metformin monotherapy or metformin in combination with insulin secretagogues at stable doses for at least 2 consecutive months at screening (a daily dose of NLT 1,500 mg or a maximum tolerated dose and NLT 1,000 mg/day for metformin, and a dose of NLT half of the maximum dose as recommended in local IFU or the maximum tolerated dose for insulin secretagogues).
4. Patients with stable living habits 2 months prior to screening, e.g., stable dietary habits and physical activities;
5. Patients with the fasting plasma glucose or fasting serum glucose at the clinical site and the fasting plasma glucose in the central laboratory of NMT 13.9 mmol/L (250 mg/dL) at screening period; with the fasting plasma glucose in the central laboratory of NMT 13.9 mmol/L (250 mg/dL) at V3;
6. Patients with the HbA1c level of NLT 7.0% and NMT 11.0% at screening in local laboratory, and with the HbA1c level of NLT 7.0% and NMT 11.0% at screening and V3 in the central laboratory;
7. Patients who were able to understand the procedures and methods of the study, willing to strictly comply with the clinical trial protocol, and voluntarily signed the informed consent form.

Exclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus, or a specific type of diabetes mellitus caused by damage to the pancreas or other disease (such as acromegaly or Cushing syndrome);
2. History of acute pancreatitis prior to screening or current history of acute or chronic pancreatitis.
3. Active gallbladder or biliary tract disease within 1 year prior to screening (active refers to the presence of associated symptoms);
4. Family or personal history of medullary thyroid cancer or multiple endocrine neoplasia type 2 (family refers to first-degree relatives by blood);
5. Individuals with a history of malignant tumors within the previous 5 years, except patients with cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
6. Decompensated cardiac dysfunction (New York Heart Association cardiac class III or IV) within 6 months prior to screening or currently;
7. Myocardial infarction, coronary artery bypass grafting, coronary stenting, hemorrhagic or ischemic stroke (except lacunar cerebral infarction), or hospitalization for unstable angina or transient ischemic attack within 6 months prior to screening;
8. Uncontrolled and severe cardiac dysrhythmia [e.g., second- or third-degree atrioventricular block, prolonged QT interval (QTc >450 ms)] within 6 months prior to screening and judged by the investigator to be unsuitable for participation in this trial;
9. Severe diabetic neuropathy within 6 months prior to screening;
10. History of diabetic foot ulcer within 1 year prior to screening;
11. Proliferative diabetic retinopathy within 6 months prior to screening or at the time of screening [confirmed by fundus photography without mydriasis or by fundus examination with medicated mydriasis (unless mydriasis is contraindicated) by an eye health care provider, or a history of laser treatment for proliferative diabetic retinopathy within 6 months prior to screening];
12. Diabetic ketoacidosis or hyperglycemic hyperosmolar state occurred within 6 months before screening to before randomization;
13. History of 2 or more episodes of severe hypoglycemia within 6 months prior to screening or severe hypoglycemia between screening and pre-randomization (see Section 3.3.2.1 of version 1.2 of the protocol for definition of hypoglycemia);
14. Previous (e.g., major or total gastrectomy, sleeve gastrectomy, gastric bypass) or current history of significant gastrointestinal disease (e.g., active ulcers, gastroparesis, pyloric obstruction, intestinal obstruction, inflammatory bowel disease, etc.) or chronic gastrastric-related surgery disease that requires long-term use of medications directly affecting gastrointestinal peristalsis and judged by the investigator to be unsuitable to participate in this trial;
15. Severe trauma or moderate to major surgery within 1 month prior to screening and up to the time of randomization or the need for systemic use of anti-infective medications and, in the judgment of the investigator, the above conditions may affect glycemic control; Prohibited treatments and/or drugs
16. Currently using weight-loss drugs, or the patient's weight has changed significantly (change NLT 10%) within 3 months before screening;
17. Received treatment with glucose-lowering medications other than metformin or insulin secretagogue (including traditional Chinese medicine with glucose-lowering effects or glucose-lowering medications under clinical validation) within 3 months prior to screening;
18. Continuous use of insulin treatment for more than 2 weeks within 1 year before screening (the time for gestational diabetes mellitus receiving insulin treatment is not within this limit);
19. Prior treatment with a dipeptidyl peptidase 4 (DPP-4) inhibitor or glucose-dependent insulinotropic polypeptide (GIP) or glucagon-like peptide-1 (GLP-1) receptor agonist and discontinuation due to lack of safety and/or efficacy;
20. Received treatment with any other investigational product or device within 3 months prior to screening;
21. Received systemic glucocorticoids (other than inhaled or topical use) or growth hormone treatment within 3 months before screening;
22. Being on warfarin at the time of screening and unable to discontinue it for the duration of the study; Laboratory findings
23. Systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg after 5 minutes of sedentary rest at screening or on the day of randomization [if the above criteria are met, the test can be repeated 2 more times (each time more than 1 minute apart) and the average of the 3 tests will be taken and judged again by the above criteria];
24. Estimated glomerular filtration rate (eGFR) <60 mL/min or urine protein qualitative test NLT ++;
25. Alanine aminotransferase (ALT) or/and aspartate aminotransferase (AST) >2.5 × ULN (upper limit of normal range) or total bilirubin level >1.5 × ULN (upper limit of normal range);
26. Currently accompanied by thyroid dysfunction that cannot be controlled with a stable drug dose (referring to a stable dose for 4 weeks or more) or abnormalities of clinical meaningfulness in thyroid function test results (TSH, FT4, FT3) during screening;
27. Currently suffering from anemia (hemoglobin level in males <120 g/L, females <110 g/L)) or other conditions that interfere with HbA1c testing;
28. Fasting triglycerides >5.64 mmol/L (500 mg/dL);
29. Serum amylase or serum lipase >3 × ULN (upper limit of normal range);
30. Hepatitis B surface antigen positive, hepatitis C antibodies positive or HIV antibodies positive (weak positive is regarded as positive); Gender and reproductive status
31. Positive pregnancy test result at screening;
32. Pregnant or lactating female at enrollment;
33. Female subjects of childbearing potential or male subjects whose sexual partner is a female of childbearing potential who are unwilling to use effective, medically approved contraception (including condoms containing sperm-inactivated spermatozoa, vaginal septum, and oral or injectable contraceptives) during the study and for 3 months after discontinuation; Other criteria
34. Alcoholics [>2 units of alcohol per day and >14 units of alcohol per week (1 unit of alcohol consumption is equivalent to 150 mL of wine or 350 mL of beer or 50 mL of spirits)] or a drug abuse history;
35. Blood donation or transfusion NLT 400 mL within 3 months prior to screening;
36. Intellectual disability or severe mental illness affecting the signing of informed consent or adherence to the study protocol;
37. Known allergies to ebenatide, human albumin (the raw material for the ebenatide formulation), empagliflozin, or related excipients;
38. Known intolerance to ebenatide or empagliflozin;
39. Other circumstances that the investigator deems inappropriate for participation in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at the end of double-blind treatment period | Week 25 visit
  The double-blind treatment period ended at the 25-week visit.

SECONDARY OUTCOMES:
Proportion of subjects with HbA1c <7.0% at the end of the double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Proportion of subjects with HbA1c <6.5% at the end of the double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting weight at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting waist circumference at the end of double-blind /open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting plasma glucose at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting proinsulin at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting insulin at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting C-peptide at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting lipids (total cholesterol) at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting lipids (low-density lipoprotein [LDL]) at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting lipids (high-density lipoprotein [HDL]) at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting lipids (triglycerides) at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting lipids (LDL/HDL ratio) at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in systolic blood pressure [SBP] at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in diastolic blood pressure [DBP] at the end of double-blind treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in 6-point finger-stick blood glucose at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in blood AST at the end of double-blind/open-label treatment period in patients diagnosed with fatty liver on screening imaging. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in blood ALT at the end of double-blind/open-label treatment period in patients diagnosed with fatty liver on screening imaging. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Change from baseline in HbA1c at the end of open-label treatment period. | Week 53 visit.
  The open-label treatment period ended at the 53-week visit.

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Prof., Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No